CLINICAL TRIAL: NCT01843829
Title: A Randomised Phase II Study of Two Pre-operative Chemoradiotherapy Regimens (Oxaliplatin and Capecitabine Followed by Radiotherapy With Either Oxaliplatin and Capecitabine or Paclitaxel and Carboplatin) for Resectable Oesophageal Cancer
Brief Title: A Feasibility Study of Chemo-radiotherapy to Treat Operable Oesophageal Cancer
Acronym: NeoSCOPE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lisette Nixon (Other Government)
Collaborators: Cancer Research UK (Other)
Responsible Party: Sponsor-Investigator, Lisette Nixon, Senior Trial Manager, Velindre NHS Trust
Organization: Velindre NHS Trust (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012/VCC/0009
Record Dates: First submitted 2013-03-07; First posted 2013-05-01 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Oesophageal Cancer
Keywords: Oesophageal cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Oxaliplatin; Capecitabine; Carboplatin; Paclitaxel; Radiotherapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carboplatin and Paclitaxel Arm (Experimental): 2 cycles OxCap: Oxaliplatin 130mg/m2 Day 1 (IV infusion) Capecitabine 625mg/m2 bd Day 1- 21 (oral)
  then CRT: Paclitaxel 50mg/m2 Days 1,8,15,22,29 (IV infusion); Carboplatin AUC 2 Days 1,8,15,22,29 (IV infusion) XRT: 45 Gy in 25 fractions
  then surgery.
  All drugs will be sourced from local stock
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Radiotherapy; Procedure: Surgery
- Oxaliplatin and Capecitabine Arm (Experimental): 2 cycles OxCap: Oxaliplatin 130mg/m2 Day 1 (IV infusion) Capecitabine 625mg/m2 bd Day 1- 21 (oral)
  then CRT: Oxaliplatin 85mg/m2 Days 1, 15, 29 (IV infusion); Capecitabine 625mg/m2 bd (oral) only on days when receiving RT XRT: 45 Gy in 25 fractions*
  then surgery.
  All drugs will be sourced from local stock
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Radiation: Radiotherapy; Procedure: Surgery

INTERVENTIONS:
Drug: Oxaliplatin
Drug: Capecitabine
Drug: Carboplatin
  Arms: Carboplatin and Paclitaxel Arm
Drug: Paclitaxel
  Arms: Carboplatin and Paclitaxel Arm
Radiation: Radiotherapy
Procedure: Surgery — Patients will have their tumour surgically removed by two-phase oesophagectomy and two-field lymphadenectomy.

SUMMARY:
About 7500 patients are diagnosed with oesophageal cancer each year in the UK of which less than a quarter have resectable disease at diagnosis. There is a general lack of consistency in the standard of care for patients across UK hospitals. Patients are either treated with a) chemotherapy followed by surgical removal of the tumour, or b) chemoradiotherapy followed by removal of the tumour by surgery, as part of their standard of care. Recent research supports the latter treatment, as chemoradiotherapy maybe more effective at shrinking the tumour and preventing the disease from spreading than taking chemotherapy alone. However, there is no definitive way of identifying which treatment is best without a clinical trial.

Evidence suggests that the effect of the chemoradiotherapy currently used as standard practice may be improved and the side effects reduced by using a different chemoradiotherapy combination. In this trial, eligible patients will receive 2 cycles of the same chemotherapy before being randomised to receive two different chemoradiotherapy regimens (carboplatin and paclitaxel verses oxaliplatin and capecitabine) both of which have shown promising results in previous studies. Patients will then have their tumour removed. The best chemoradiotherapy regimen will then be taken forward to a Phase III trial in which chemoradiotherapy will be compared with chemotherapy alone.

The efficacy of the regimens will be measured by counting the number of patients who i) remain free from cancer, ii)have local or distant spread of their cancer, iii) are successfully recruited and iv) experience toxicities. A specific set of toxicity criteria will be used to monitor any treatment induced side-effects and provide justification for any necessary dose modifications or withdrawal of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed operable oesophageal cancer (adenocarcinoma)
* Tumour must be staged as a T3, 4 or N1 (using TNM6 staging) or T3, T4a or N13 using TNM7 staging)
* Maximum disease (Tumour plus nodes) length 8 cm staged with EUS and CT/PET
* WHO performance status 01
* Adequate haematological, renal, respiratory, cardiac and hepatic function
* The patient has provided written informed consent.

Exclusion Criteria:

* Histologically confirmed operable oesophageal cancer (squamous cell carcinoma)
* Uncontrolled angina pectoris, myocardial infarction within 6 months, heart failure, clinically significant uncontrolled cardiac arrhythmias, or any patient with a clinically significant abnormal ECG.
* Patients with any previous treatment for oesophageal carcinoma.
* Siewert type 3 oesophagogastric tumours.
* T4 tumours invading contiguous structures other than diaphragm, crura or mediastinal pleura.
* Patients with disease in any of the following areas on the CT scan, EUS or other staging investigation:

  1. Evidence of metastases in liver, lung, bone or other distant metastases.
  2. Abdominal para aortic lymphadenopathy >1cm diameter on CT or >6mm diameter on EUS.
  3. Invasion of tracheo-bronchial tree, aorta, pericardium or lung.
* Lymphadenopathy encasing the coeliac axis (as described above, patients with single nodes lying anterior to the origin of the splenic artery and anterior to the origin of the coeliac axis are not excluded).
* Any patient with a single significant medical condition which is thought likely to compromise his or her ability to tolerate any of the above therapies.
* Specific contraindications to surgery, chemotherapeutic agents (including known allergies to chemotherapy) or radiotherapy.
* Pregnant or lactating women and fertile women who will not be using adequate contraception during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy | 24 months
  The efficacy of the trial treatment will be assessed by conducting analysis on the resected tumour specimen of participants undergoing surgery. This will be achieved by looking at the pathological complete response rate (pCR).

SECONDARY OUTCOMES:
Feasibility of recruiting 62 patients within 18 months | 18 months
  Feasibility of recruiting to a pre-operative chemoradiotherapy trial in the UK will be determined by recruitment within 18 months.
Safety | 3 years
  The trial safety will be assessed by looking at the toxicity. Toxicities during treatment and at 6 and 12 months post-surgery will be recorded using the CTCAE version 4. SAEs will be collected in real time. The morbidity/mortality rate post surgery will also be assessed.
Efficacy | 5 years
  The efficacy will be measured as a secondary end point by assessing the median, 3 and 5 year overall survival.
Efficacy | 24 months
  The CRM (circumferential resection margin) which is a measurement of how successful the surgery was in removing all traces of tumour, will be assessed.

CONTACTS AND LOCATIONS:
Locations (12):
- United Kingdom (12):
  - Bristol Oncology and Haematology Centre, Bristol
  - Valindre NHS, Cardiff
  - University Hospitals Coventry and Warwickshire, Coventry
  - Royal Derby Hospital, Derby
  - St James's Hospital, Leeds
  - Leicester Royal Infirmary, Leicester
  - St Mary's Hopsital, London
  - The Christie, Manchester
  - Churchill Hospital, Oxford
  - Weston Park Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - The Great Western Hospital, Swindon

REFERENCES:
- [Derived] Mukherjee S, Hurt C, Radhakrishna G, Gwynne S, Bateman A, Gollins S, Hawkins MA, Canham J, Grabsch HI, Falk S, Sharma RA, Ray R, Roy R, Cox C, Maynard N, Nixon L, Sebag-Montefiore DJ, Maughan T, Griffiths GO, Crosby TDL. Oxaliplatin/capecitabine or carboplatin/paclitaxel-based preoperative chemoradiation for resectable oesophageal adenocarcinoma (NeoSCOPE): Long-term results of a randomised controlled trial. Eur J Cancer. 2021 Aug;153:153-161. doi: 10.1016/j.ejca.2021.05.020. Epub 2021 Jun 20. PMID 34157617
- [Derived] Mukherjee S, Hurt CN, Gwynne S, Sebag-Montefiore D, Radhakrishna G, Gollins S, Hawkins M, Grabsch HI, Jones G, Falk S, Sharma R, Bateman A, Roy R, Ray R, Canham J, Griffiths G, Maughan T, Crosby T. NEOSCOPE: A randomised phase II study of induction chemotherapy followed by oxaliplatin/capecitabine or carboplatin/paclitaxel based pre-operative chemoradiation for resectable oesophageal adenocarcinoma. Eur J Cancer. 2017 Mar;74:38-46. doi: 10.1016/j.ejca.2016.11.031. Epub 2017 Feb 8. PMID 28335886
- [Derived] Mukherjee S, Hurt CN, Gwynne S, Bateman A, Gollins S, Radhakrishna G, Hawkins M, Canham J, Lewis W, Grabsch HI, Sharma RA, Wade W, Maggs R, Tranter B, Roberts A, Sebag-Montefiore D, Maughan T, Griffiths G, Crosby T. NEOSCOPE: a randomised Phase II study of induction chemotherapy followed by either oxaliplatin/capecitabine or paclitaxel/carboplatin based chemoradiation as pre-operative regimen for resectable oesophageal adenocarcinoma. BMC Cancer. 2015 Feb 12;15:48. doi: 10.1186/s12885-015-1062-y. PMID 25880814